CLINICAL TRIAL: NCT02919215
Title: Teacher Help: Novel Technologies for Meeting the Immediate Needs of Youth With Mental Health Disorders in Canada
Brief Title: Teacher Help for Children and Youth With Mental Health Disorders
Acronym: TeacherHelp
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There were many challenges with recruiting participants. Since we had fewer participants than expected complete baseline procedures, the research team changed the study design to a pre-post design. Therefore, no participants were enrolled in the RCT.
Sponsor: IWK Health Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 143552
Record Dates: First submitted 2016-09-22; First posted 2016-09-29 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2019-08

CONDITIONS: Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder; Learning Disabilities
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Teacher Help Intervention (Experimental): The intervention will be provided to collaborating psychologists and their teachers to access. Teachers will work through the intervention, and psychologists will act as a support for teachers if needed. All participants can access and/or provide usual services. Teachers will work with one student in their classroom with ADHD, ASD, or LD throughout the intervention phase. Each session in the program will provide factual information to teachers, strategies for implementation of best practices to address the specific mental health disorder in the classroom setting (i.e., ADHD, ASD, or LD), and access to additional help and advice.
  Interventions: Behavioral: Teacher Help Intervention

INTERVENTIONS:
Behavioral: Teacher Help Intervention — The intervention will be provided to collaborating psychologists and their teachers to access. Teachers will work through the intervention, and psychologists will act as a support for teachers if needed. All participants can access and/or provide usual services. Teachers will work with one student in their classroom with ADHD, ASD, or LD throughout the intervention phase. Each session in the program will provide factual information to teachers, strategies for implementation of best practices to address the specific mental health disorder in the classroom setting (i.e., ADHD, ASD, or LD), and access to additional help and advice.

SUMMARY:
Currently, Canadian school systems are struggling to meet the needs of children with mental health disorders. It is particularly challenging to meet the needs of students with neurodevelopmental disorders (NDDs) within the regular classroom setting. Past research indicates that supportive and knowledgeable teachers who implement evidence-based interventions in the classroom are effective in increasing the success of students with mental health disorders, including students with NDDs. Factors such as understanding the disorder, use of evidenced-based teaching approaches, and access to professional developmental opportunities can improve teacher's knowledge and classroom practice. The Teacher Help research team along with industry partner, Velsoft, and key knowledge user, Nova Scotia Department of Education and Early Childhood Development, will address this need by developing, evaluating, and commercializing a sustainable eHealth resource for teachers. Teacher Help is an eHealth professional development program that assists teachers who work in the regular classroom setting in providing evidence-based interventions to students in grades 1 to 12 with mental health disorders. The program was developed based on programs previously tested by the investigators as well as on the extant literature on this topic. Teacher Help provides access to information through 6 sessions using text, video, and activities. Currently three modules (Attention-Deficit/Hyperactivity Disorder [ADHD], Autism Spectrum Disorder [ASD], and Learning Disabilities [LD]) are at different stages in the innovation pipeline.Our goal is to conduct a pre-post intervention study in which participants (collaborating school psychologists, teachers, students, and caregivers) access the Teacher Help program. The effects of the Teacher Help intervention will be assessed once participants have completed the intervention. Assessments will include students' general psychopathology symptoms, impairment, and quality of life as reported by teachers, parents/caregivers, and students (when developmentally appropriate). Additionally, we will explore changes in treatment utilization, participants' satisfaction with the program, as well as changes in teachers' beliefs toward students with NDDs and use of evidence-based strategies. To the Teacher Help team's knowledge, Teacher Help is the first and only research-validated eHealth program directly targeting teachers to help them intervene with children and youth who have mental health disorders, thus allowing Canada to take a lead in eHealth as applied to a school context.

DETAILED DESCRIPTION:
The current research study will evaluate the effectiveness of an eHealth professional development program, Teacher Help, that assists teachers in understanding mental health disorders and providing evidence-based interventions to students in grades 1 to 12 with mental health disorders. If effective, we will work with our partners to commercialize this program for a reasonable rate, so that all school boards in Canada can have access to this intervention.

The primary objective is to assess the impact (baseline vs. 2

-month follow-up) of the intervention on students' symptoms of general psychopathology as reported by teachers.

The secondary objectives are to: a) assess the difference in impact (baseline vs. 2-month follow-up) on students' general psychopathology as reported by teachers across the three diagnostic groups (i.e., ADHD, LD, and ASD), b) evaluate the impact (baseline vs. 2-month follow-up) of the intervention on teacher ratings of student impairment, c) evaluate the impact (baseline vs. 2-month follow-up) of the intervention on teacher ratings of the students' quality of life, d) assess participants' satisfaction with the Teacher Help program, and e) determine if the effects are noticeable by parents/caregivers (here after referred to as parents).

Exploratory research objectives include whether the following variables following the intervention: a) teachers' belief systems toward students with ADHD, ASD, and LD, b) teachers' use of evidence-based interventions, and c) students' perceptions of their level of general psychopathology, impairment, and quality of life. We will also determine whether: d) demographic characteristics (e.g., student's grade, teachers age and experiences) are related to outcome, e) process-level changes are evident across the intervention sessions, f) teachers' use of Teacher Help influences treatment utilization outside of the Teacher Help program, and g) satisfaction is related to willingness to pay for the program.

The Teacher Help intervention is an online professional development program designed to increase classroom teachers' knowledge about NDDs and to assist them in providing evidence-based interventions to students in grades 1 to 12 in the regular classroom setting. Grade primary/kindergarten is not included due to the transitional nature of this first year of formal education. Evidenced-based strategies are incorporated throughout the intervention, such as reward programs for students with ADHD, functional behaviour programs for students with ASD, and appropriate adaptations and remediation for students with LD. The program is designed to be self-guided; however, teachers are encouraged to collaborate with their school teams (e.g., school psychologists, resource teachers) throughout the program.

The intervention is delivered via Velsoft® Training Materials eLearning platform Znanja, which delivers through participants' desktops, laptops, tablets, and smartphones the interactive, guided interventions, and strategies that can be used in the classroom. The Teacher Help program supports the use of evidenced-based techniques in the classroom, through combining graphics, interactive elements, and video to engage and encourage teachers. The program can be used at a time that is convenient for teachers, removing access barriers and providing services to students with mental health disorders.

Each module (ADHD, ASD, LD) includes six sessions made available sequentially to participants. Each module includes the following session topics: 1) An evidence-derived overview of the disorder and its treatments; 2) How teachers can help and the team approach; 3) The main intervention focused on core symptoms and how to implement this in the classroom; 4) Additional classroom strategies that may be helpful in addressing the core symptoms of the disorder; 5) Additional needs of individuals in relation to common comorbid symptoms and how to help; 6) Wrapping up the program and planning for the future.

The sessions are made available to teachers one per week; however, teachers can spend up to two weeks on each session, if they so choose. As such, the completion time of the intervention will range from 6 - 8 weeks. Each session will provide evidence-based information to teachers, strategies for implementation of best practices to address the specific mental health disorder in the classroom setting and will encourage teachers to reach out to the school team for additional help and advice. Teacher Help can be individualised and is designed to be flexible and adaptable to fit the needs of the student and the teacher.

The Project Coordinator will provide teachers with login information to Teacher Help. School psychologists will be provided with a manual outlining the philosophy and technical aspects of the Teacher Help program and will verify that the program is a good fit for the student the teacher wishes to work with (and may in fact help the teacher to select an appropriate student to work with). Once teachers have access to the program, they are encouraged to communicate and collaborate with their school team, including their school psychologist, school administrators, specialized teachers, and other classroom teachers, through usual communication channels (e.g., school email, face-to-face meetings), for support with implementing the Teacher Help program.

Over the past 10 years, several research studies have taken place to evaluate and test the Teacher Help program. In 2006, a research team and educator team collaborated to better understand teachers' professional development needs when working with students with autism spectrum disorder (ASD). Teachers consistently emphasized the need to be able to access professional development resources that have been vetted and organized by experts, so they can trust that the suggestions are evidence-based and can follow a well-laid out plan as needs arise. Applying the eHealth concept seemed a promising solution to the barriers teachers face in mental health professional development. The information learned from this study was applied to ADHD as the first experiment with an eHealth solution.

A usability study of the Teacher Help for ADHD module took place in 2010 to test whether a web-based platform would be an effective tool for supporting knowledge, attitude, and behavior change in teachers of elementary school children with ADHD. Results revealed that teachers' knowledge positively changed from pre- to post-intervention, as did teachers' attitudes related to perceived control in their classrooms, and sense of competence in teaching. Teachers expressed that they would have liked to have someone to consult with while using the program both in private messaging and on a Discussion Board. As such the subsequent randomized controlled trial (RCT) testing the effectiveness of the Teacher Help for ADHD module included access to a psychologist who was called the ADHD Coach through an online Discussion Board and private e-messaging.

From 2012 - 2013, 58 elementary classroom teachers in Nova Scotia, Canada, along with their students with ADHD, participated in a RCT to test the effectiveness of the Teacher Help for ADHD module. Online questionnaire data was collected from teachers and parents pre-intervention, post-intervention (6 weeks), and after an additional 6-week follow-up. Intent-to-treat analyses found significant improvements based on teacher (but not parent) reports of core ADHD symptoms and impairment for the Intervention group relative to the control group. Ratings of ADHD symptoms using the Connors 3 ADHD Index T-score demonstrated a statistically significant and clinically relevant change in scores for the Intervention group at both the 6-week and 8-week assessment points. Satisfaction ratings for the content of the intervention were all above 84%, while ratings for the Discussion Board and Coaching aspects of the program received a satisfaction rating of 70%. Participants engaged in almost all the intervention components (i.e., session content, worksheets, and supplemental materials); however, they did not fully engage in the Discussion Board and Coaching aspects of the program (e.g., approximately 14% of teachers accessed the Coach). It was concluded that Teacher Help is a feasible, acceptable, and effective intervention.

In 2013 a usability study took place to evaluate the content in the Elementary School version of the Teacher Help for LD module. Led by Ashton Parker (Masters of School Psychology student at Mount Saint Vincent University [MSVU]), under the supervision of Dr. Penny Corkum, Dr. Melissa McGonnell (Associate Professor at MSVU), and Annie Baert (Learning Disabilities Consultant at Nova Scotia Department of Education and Early Childhood Development), the study was conducted with a prototype of the Teacher Help for LD module, and both qualitative and quantitative data were collected. Nineteen experts on learning disabilities (e.g., school psychologists, resource teachers) reviewed the intervention and provided an overall satisfaction rating of 4.37 out of 5. Results from this study were used to revise the Teacher Help for LD module to finalize content.

To date, the Teacher Help for ASD module has not undergone usability testing. However, usability testing of the Teacher Help for ASD module will occur prior to completing the cluster randomized controlled trial of this module. We will conduct usability testing in Nova Scotia (NS) using methodology we have used in previous research. The module will be revised based on the usability study results, and these will be incorporated into the online program. An ethics application for this study was submitted to the IWK Health Centre Research Ethics Board (REB) on Monday, February 27th, 2017.

Previous versions of the Teacher Help program were delivered via Dalhousie University's learning management system BBLearn; however, this system is limited and cannot be commercialized. As such, we needed to move to a platform that would allow for larger clustered randomized controlled trails (RCTs) and for eventual commercialization. In February to April 2016 a usability study was conducted, funded by Springboard Atlantic, to evaluate user experience and satisfaction with Velsoft® Training Materials' eLearning platform Znanja using a prototype of the Elementary School version of the Teacher Help for ADHD module. The content was not the focus of this review given that it had been reviewed previously. Participants indicated that they liked the look and feel of the platform (e.g., colours were calming and not too overwhelming), that the program could be navigated with ease, and that they liked that they were able to track their progress through each of the sessions. Participants indicated that it would be helpful to have the worksheets available for downloading in multiple spots throughout the program and that more pictures would be ideal. These results have been used to revise components of the online Teacher Help program. As a method of ensuring that all users are able to navigate the program with ease, a video tutorial will be provided to users for review once they have been given access to the Teacher Help program.

The study is a pre-post intervention study. CONSORT 2010 guidelines and CONSORT eHealth guidelines were used to design the trial and will be adhered to when reporting the trial.

The study will recruit participants from across Canada. The study will be coordinated through Corkum LABS at Dalhousie University. Collaborating school psychologists will be asked to recruit a minimum of 6 to a maximum of 12 teacher-student-parent triads (we will ask school psychologists to commit to recruiting a maximum of 12 interested teachers, but we will need to flexible with this criterion in order to accommodate the different roles and demands of school psychologists). We will try to recruit school boards from each of the 5 Canadian regions: Atlantic Region, Central Canada, Prairie Provinces, West Coast, and North. All participants will be able to access standard care (i.e., all available resources and additional programs and services available to them) while enrolled in the study.

The Teacher Help program involves minimal risk to the participants. Participants are provided with the email address of the Project Coordinator and the Principal Investigator who they may contact in the event that they have concerns or questions related to the study.

The study safety monitoring plan involves a 3-step process. First the Project Coordinator, who will be in contact with participants as they complete the battery of assessments, will communicate with the Principal Investigator of this study, Dr. Penny Corkum, a registered psychologist, any difficulties experienced by the participants that cannot be dealt with by the trained Project Coordinator (who is trained as a school psychologist). Any difficulties will be immediately communicated to Dr. Corkum or her delegate (always a registered health care provider), and follow-up with the participant will be made to ensure their well-being. The second step would be enacted if Dr. Corkum determined that she needed further consultation to address the concern raised by a participant. She would communicate with the co-investigators, which includes 2 psychologists and 1 psychiatrist, who have expertise in all three NDDs. The third step would be enacted if: resolution was not achieved at step 2, if there are differences of opinions among the investigators, or if an adverse event did happen. The third step involves communication with an arms-length Safety and Adverse Events Committee, which we will be comprised of four members of the Teacher Help advisory counsel not directly associated with the day-to-day implementation of the Teacher Help research study, who will represent school psychologists, educators, parents, and youth with NDDs, who will review the problem and provide their advice, which will be followed by the research team.

Participants will be recruited from across all Canadian provinces and territories. Inclusion and Exclusion criteria are different depending on participant group (e.g., collaborating school psychologists, teachers, students, and parents). All participants need to have regular access to high-speed internet connection and an email account, as well as be willing to participate in research.

The recruitment strategy for this study will be broadly based across Canada using a multi-prong approach targeting four groups: 1) school boards, 2) school psychologists, 3) external stakeholders and organizations (i.e., our partners including healthcare provider associations), and 4) the media.

The target audience of the Teacher Help intervention is school psychologists working within school systems with regular access to the internet. Therefore, the recruitment strategy will be primarily based on online tools, most notably the study website. Social media will also be used; for example, Facebook and Twitter. Traditional recruitment methods will also be employed, including sharing of information sheets and conference presentations, to reach both potential participants and the education community.

The pre-screening process is complex as it requires ongoing communication with the collaborating school psychologist in the school and other relevant school personnel. Each province and each school board can have different criteria for engagement with research. We will first ensure that the school board meets our criteria for participating through an online screening process. Interested school psychologists and/or school personnel that represent the school board will first be asked to sign a Screening Information and Consent Form detailing the screening process. Once the consent process if complete, the participant will be asked to complete the online screening questionnaire which asks for information about their school board such as location, size, and requirements for completing research within the school board.If the school board meets screening criteria, we will then begin the process of navigating the school board's system in terms of permissions needed to complete research. This will most often require the approval of those that supervise participating school psychologists as well as approval from the school board and schools for participation in research; for some school boards this is a full ethics review process, for other school boards this is sharing our ethics approval from IWK, and for others it may just be approval without any review process. For those School Boards that require a review, we will help facilitate this process by completing any necessary applications and providing appropriate documentation of ethical clearance from the IWK Health Centre as needed.

School psychologists will consent to participate in the study by completing the Information and Consent Form for Collaborating School Psychologists. School psychologists will be given the opportunity to contact the Project Coordinator by email to have questions answered and concerns addressed. It is important to note that typically the school psychologist will have had ongoing communication with the Project Coordinator and investigators up to this point and will have had ample opportunity to ask questions about the study.

After the school board and schools have given their approval for participation in the study and once the collaborating school psychologist agrees to participate in the study, collaborating school psychologists will be asked to approach teachers about participating. Collaborating school psychologists will be asked to work with the teachers to identify potential students who fit the criteria of the research study and would potentially benefit from the program. As part of this process, the collaborating school psychologist will review the identified student's file to confirm their diagnosis of ADHD, ASD, or LD. The collaborating school psychologist will have been provided with all informational materials to help with recruitment of teacher-student-parent triads. The goal is for each collaborating school psychologist to recruit a minimum of 6 to a maximum of 12 teachers. Once a teacher has identified a potential student, the collaborating school psychologist will send the teacher a link to an online consent form for the teacher to sign electronically. Once a teacher consents, he/she will send an email to the student's parents asking for their consent to work with their child using the Teacher Help program. Once consent is gained from the parent by completing the online consent form, the collaborating school psychologist will approach the student to gain their assent. The collaborating school psychologist will review information about the study with the student and electronically sign a form to indicate that she/he has reviewed the information and has answered all the student's questions. All participants will be given the opportunity to contact the Project Coordinator and Principal Investigator by email or phone to have questions answered and concerns addressed. The Project Coordinator will notify collaborating school psychologists as teacher-student-parent triads complete the consent process.

Eligible school psychologists, teachers, and parents will be asked to provide their email address and phone number when completing their Information and Consent Forms. This will enable the researchers to send the baseline and follow-up measures as well as reminders to complete these measures electronically via REDCap.

Outcome measures will be completed by collaborating school psychologists, teachers, parents, and students (when developmentally appropriate) at baseline, and follow-up assessments at 2--month post-randomization. . All measures will be administered using the REDCap database.

Each teacher will complete 1 module (i.e., ADHD, ASD, or LD) to address the needs of the student who they identified to participate in the study. Teachers will complete the six sessions of the Teacher Help program which includes reviewing session information, completing worksheets and activities, accessing supplemental materials if they so choose, and implementing the classroom strategies outlined in the program. Prior to each session of the intervention, teachers will be asked to complete a short questionnaire asking about their students' level of impairment before beginning the session. This is so we can perform a process analysis across the sessions. Teachers can access other services, outside of Teacher Help, as usual.

Notes for teachers of students in High School: Many high schools have a semester system (e.g., Fall and Winter Semesters); as such, it is possible that the student a teacher chooses to work with in the beginning of the school year will not be in that same teacher's class once the semester changes. In the event that this occurs, it will be essential that the teacher participating in the study finds an alternative teacher, who is currently teaching the student, to continue to implement the Teacher Help program with the student. In order to maintain consistency, we ask that the teacher who initially began the program with their student completes the questionnaires collaboratively with the new teacher for any follow-up assessments.

Collaborating school psychologists will be provided with a manual outlining their role and expectations within the Teacher Help program. School psychologists will be available for collaboration through usual communication channels (e.g., school email, face-to-face meetings) if teachers have questions about or need support with implementing the Teacher Help program. They are allowed to provide other services, outside of Teacher Help, as usual.

ELIGIBILITY:
Potential school psychologists must meet the following criteria to be eligible to participate in this study:

1. Are licenced/registered psychologists OR are psychological associates OR are certified school psychologists OR are on the candidate register
2. Work within or for a public-school system within Canada
3. Have the ability to recruit a minimum of 6 to a maximum of 12 classroom teachers who teach grades 1-12 to participate (some flexibility available). A student of each teacher and his/her parents need to agree to participate as well.
4. Willing to provide support to teachers during the implementation of the Teacher Help program (approximate maximum of 30 minutes/week overall)

Exclusion Criteria for Collaborating School Psychologists

Potential psychologists who meet any of the following criteria are not eligible to participate in the study:

1. Are planning to be on a leave of absence at any time during the duration of the study
2. Work within a school system where there is no English instruction

Inclusion Criteria for Teachers

Potential teachers must meet the following criteria to be eligible to participate in this study:

1. Work in a regular classroom setting in the public-school system in grades 1-12 with English as the language of instruction
2. Currently have one student in their classroom with ADHD, LD, or ASD who they would like to help by using this program
3. The parent and student have agreed to participate

Exclusion Criteria for Teachers

Potential teachers who meet any of the following criteria are not eligible to participate in the study:

1. The teacher participated in any of the previous Teacher Help studies
2. Plan to be on a leave of absence at any time during the duration of this study

Inclusion Criteria for Families (i.e., parents and students)

Potential families (i.e., parents and students) must meet the following criteria to be eligible for this study. Specifically, we are looking for families where:

1. The child attends public school in the English stream grades 1 to 12
2. The child has been diagnosed with ADHD, LD or ASD.

   a. For students with ADHD or ASD, the child will need to have been diagnosed by a physician or psychologist. For students with LD, the child will need to have been diagnosed by a psychologist. Documentation on the student's file should indicate this diagnosis. We will not ask for this documentation, but request that the collaborating school psychologist confirms that this documentation exists and to indicate when the diagnosis was made and by what type of health professional (e.g., physician, psychologist)
3. The child spends at least two-thirds of their class time inside the typical classroom (i.e., no more than one-third of class time is spent in a special education setting)
4. The student is either on a stable dose of medication for the specific NDD or no medication with no plan to start/change medication for the next 5 months

Exclusion Criteria for Families (i.e., parents and students)

Potential families that meet any of the following criteria are not eligible to participate in the study. Specifically, families where:

1. The student's primary diagnosis is not ADHD, LD, or ASD (i.e., it is not the diagnosis that is causing the most negative impact in the school context)
2. The student is on an Individualized Program Plan (IPP)/Individual Education Plan (IEP) and/or Alternative Program Plan due to significant physical, behavioural, communication, or cognitive difficulties and as such require significant teaching/educational assistant involvement or time spent in specialized learning environments

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ; Goodman, 2001) | Baseline, Follow Up
  The SDQ will be used to measure student behavior using a Likert Scale with three possible choices ranging from "Not True" to "Somewhat True" to "Certainly True". "Somewhat True" is always scored as 1, but the scoring for "Not True" and "Certainly True" varies with the item (either scored as 0 or 2), so reverse scoring will be conducted. The SDQ is a validated, 25-item modular tool designed to measure student behavior. The SDQ assesses student behavior across 5 domains: emotion symptoms, conduct problems, inattention/hyperactivity, social problems and prosocial behaviour. The total difficulties score is generated by summing scores of all scales except the prosocial scale, resulting in a range of 0-40. The scores are transformed to a 0-10 scale, with higher scores reflecting more negative interference in the child's life. Higher prosocial scale scores indicate more prosocial behavior.

SECONDARY OUTCOMES:
Teacher Demographic Questionnaire (author made) | Baseline
  A 18-item questionnaire completed by teachers. Queries age, sex, years of experience as a teacher, number of youth taught with the disorder of interest (i.e., ADHD, ASD, LD), and perceived knowledge of the disorder rated on a 5-point scale ranging from 0 (No knowledge) to 4 (Very knowledgeable). These data will be used to describe the sample.
Parent Demographic Questionnaire (author-made) | Baseline
  A 16-item questionnaire to be completed by parents. Will be used to collect information to describe the sample (e.g., family income, ethnicity, marital status).
Collaborating School Psychologist Demographic Questionnaire (CPDQ) | Baseline
  The CPDQ will be used at baseline only to collect demographic information about the collaborating psychologists. Thirty-one (31) items for this questionnaire were compiled from the previous Teacher Help for ADHD randomized controlled trial (RCT) Teacher Demographic Questionnaire.
Rating Scale of Impairment (RSI) (Goldstein & Naglieri, 2016) | Baseline, Follow Up
  The RSI was developed by Dr. Sam Goldstein and Dr. Jack Naglieri in 2016, and is a behavior rating scale that measures functional impairment across six life areas in children and youth: school/work, social, mobility, domestic, family, and self-care. A Total Score is also produced which indicates the child/youth's overall impairment. The number of items on the RSI varies depending on which form is used (Parent Form [5-12 Years] has 41 items, Parent Form [13-18 Years] has 49 items, and the Teacher Forms have 29 items). Items are rated on a 6-point likert scale from "1 - Never" to "6 - Always". An elevated T-score of 65 or above is evidence of impairment. Defining a clinical level of impairment with the RSI scores can be used to meet impairment criteria required for DSM-5 diagnostic thresholds.
  Parent and Teacher forms are available, and the questionnaire takes approximately 10 minutes to complete.
KIDSCREEN Questionnaire (KIDSQ) | Baseline, Follow Up
  The KIDSQ assess children/adolescents' subjective health and well-being. The questionnaire can be administrated in hospitals, medical establishments and schools by professionals in the fields of public health, epidemiology, and medicine (for clinical and research purposes). It is applicable for healthy and chronically ill children and adolescents from 8 to 18 years and can be completed by the children themselves. A proxy measure for parents or primary caregivers (e.g., teachers) who have day-to-day involvement with the child in question is also available. The questionnaires can be completed in person at home, in a classroom, and in other settings.
Teacher Satisfaction Questionnaire (TSQ) | Follow Up
  The questionnaire asks teachers to indicate their level of agreement on a scale of 1 (Strongly Disagree) to 6 (Strongly Agree) with each of the statements about the Teacher Help program they participated in. Questions ask about ease of completing the questionnaires, the content of the intervention, improvements in their student's behavior and academics, as well as their overall experiences with the program. The questionnaire takes approximately 5 minutes to complete.
Collaborating School Psychologist Satisfaction Questionnaire (CPSQ) | Follow Up
  The questionnaire asks collaborating school psychologists to indicate their level of agreement on a scale of 1 (Strongly Disagree) to 6 (Strongly Agree) with each of the statements about the Teacher Help program. Questions ask about ease of completing the questionnaires, the content of the intervention, improvements in student's behavior and academics, improvements in teachers use of evidence-based interventions, as well as their overall experiences with the program. The questionnaire takes approximately 5 minutes to complete.
Youth Satisfaction Measure (author-made) | Follow Up
  A 4-item questionnaire to be completed by youth when appropriate. Will assess the youth's view of the helpfulness of the program.
Parent Satisfaction Questionnaire (PSQ) | Follow Up
  The questionnaire asks parents to indicate their level of agreement on a scale of 1 (Strongly Disagree) to 6 (Strongly Agree) with each of the statements about the Teacher Help program their child participated in. Questions ask about ease of completing the questionnaires, inclusion in the school-based intervention, improvements in their child's behavior and academics, as well as their overall experiences with the program. The questionnaire takes approximately 5 minutes to complete.
Collaborating Psychologist Support Log (author-made) | Baseline, Follow Up
  The questionnaire asks the collaborating school psychologist to provide information on how often they provided support to the teacher, how they communicated with the teacher, how long they typically spent supporting the teacher, as well as area they provided support on. At 3-month follow-up school psychologists in the Intervention group are also asked to comment on any supports provided to teachers specific to the Teacher Help program. The questionnaire takes approximately 5 minutes to complete for each teacher.
Teacher Beliefs Questionnaires (TBQ) | Baseline, Follow Up
  The TBQ is an 18-tem questionnaire that will be used to assess whether the Teacher Help program was effective in improving teachers' belief systems toward students with the disorder of interest. The measure looks at 7 constructs: Lack of Control, Negative Classroom Effects, Diagnostic Legitimacy, Perceived Confidence, Influences to Management, Expectations, and External Control. However, we will be focusing only on 4 of the constructs for the purposes of this research study: Lack of Control, Negative Classroom Effects, Diagnostic Legitimacy, and Perceived Confidence.
Willingness to Pay Questionnaire (WPQ) | Follow Up
  The WPQ questionnaire is a brief author-made questionnaire that will be used to assess how valuable teachers feel the Teacher Help intervention was by asking how much participants would be willing to pay for the intervention. It also asks about what teachers and collaborating school psychologists would be willing to pay for different, but related resources. This will aid the Teacher Help investigators in understanding the potential to commercialize the program and offer additional resources as needed. The WP is only administered to those teachers and collaborating school psychologists in the Intervention group at 3 month follow-up and will consists of 3-items. The WP takes approximately 5 minutes to complete.
Treatment Utilization Questionnaire for Parents (TUQ - P) | Baseline, Follow Up
  The TUQ - P questionnaire is author made, and will be used to measure the extent to which parents utilize treatment resources (e.g., family physicians). This will be used to determine if the Intervention or Waitlist group received more/less treatment outside of the Teacher Help program. The TUQ - P includes 5 items that ask about what supports parents accessed for their child's neurodevelopmental disorder (NDD) and/or NDD related problems. The TUQ - P will be administered at the baseline, 3- and 5-month follow-up. The TUQ - P requires approximately 5 minutes to complete.
Treatment Utilization Questionnaire for Teachers (TUQ - T) | Baseline, Follow Up
  The TUQ - T questionnaire is author made, and will be used to measure the extent to which teachers utilize resources to support their student (e.g., the school psychologist). This will be used to determine if the Intervention or Waitlist group received more/less treatment outside of the Teacher Help program. The TUQ - T includes 3 items that ask about what supports were accessed for their student's neurodevelopmental disorder (NDD) and/or NDD related problems. The TUQ - T will be administered at the baseline, 3- and 5-month follow-up. The TUQ - T requires approximately 5 minutes to complete.
Impairment Rating Scale (IRS) | At the beginning of each Teacher Help section
  The IRS assesses functioning across different areas of functioning: peer, sibling, parent, teacher, academics, self-esteem, classroom/family, and globally. The IRS is sensitive to changes in behavior modification and can be used to monitor improvements.
  The IRS includes 7-items that include a 7-point scale that ranges from "0 - No problem; definitely does not need treatment or special services" to "6 - Extreme Problem; definitely needs treatment or special services" along with opportunity to provide elaborations and comments. The teacher version of the IRS is being collected as a process measure and as such will be administered before each Teacher Help session. The IRS requires approximately 10 minutes to complete.
Instructional and Behaviour Management Approaches Survey (IBMAS) | Baseline, Follow Up
  Teachers are asked to rate the frequency with which they utilize a range of instructional and behaviour management practices to manage and support students with "attention and/or behaviour problems" in the classroom. Teachers rate the frequency with which they used the various approaches on a five-point scale ranging from 1 (rarely) to 5 (most of the time). The mid-point reflected ''occasional use'' (coded as 3). A total score for the behavior management items and the instructional supports/strategies was created by summing the items within each category. The questionnaire takes approximately 5 minutes to complete.

OTHER OUTCOMES:
Screening Questionnaire (SQ) (author made) | Screening, pre-baseline
  The SQ will be used to collect information about school boards such as their size, location, and research review process before completing the consent process. This information will help the researchers to determine if a school board is eligible to participate in the Teacher Help study. The SQ requires approximately 5 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Penny V Corkum, PhD, Principal Investigator — Dalhousie University
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available. The team will engage in usual end-of-study knowledge translation, such as presenting at local, national and international conferences, as well as preparing manuscripts for high-impact open journals. We will also prepare a number of social media products (e.g., webinars) that share the results of the study. We will include the voices of our end-users in these materials; however, they will not be identified.